CLINICAL TRIAL: NCT04866212
Title: Comparison of Hand Skills, Visual-Motor Integration and Participation in Activities of Daily Living of Children With and Without Type 1 Diabetes
Brief Title: Comparison of Manual Skills, Visual-Motor Integration and Participation of Children With and Without Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, mehtap kilicoz, Msc student, Istanbul Medipol University Hospital
Other Study IDs: 10840098-604.01.01-E.14675
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes; Hand Skills; Visual Motor Integration; Participation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Type 1 Diabetes Group: Children with type 1 diabetes were evaluated in terms of their hand skills, visual motor integration, participation in daily life activities and academic success.
  Hand skills were evaluated using the Jebsen Taylor Hand Function Test. Participation was evaluated with Participation and Environment Measurement-Children and Youth. Visual motor integration was evaluated with Beery-Buktenica Developmental Test of Visual Motor Integration. Academic success was evaluated with the course success score.
  Interventions: Behavioral: Beery- Buktenica Developmental Test of Visual Motor Integration; Behavioral: Jebsen Taylor Hand Function Test; Diagnostic Test: Participation and Environment Measure - Children and Youth
- Children without Type 1 Diabetes Group: Children without type 1 diabetes were evaluated in terms of their hand skills, visual motor integration, participation in daily life activities and academic success.
  Hand skills were evaluated using the Jebsen Taylor Hand Function Test. Participation was evaluated with Participation and Environment Measurement-Children and Youth. Visual motor integration was evaluated with Beery-Buktenica Developmental Test of Visual Motor Integration. Academic success was evaluated with the course success score.
  Interventions: Behavioral: Beery- Buktenica Developmental Test of Visual Motor Integration; Behavioral: Jebsen Taylor Hand Function Test; Diagnostic Test: Participation and Environment Measure - Children and Youth

INTERVENTIONS:
Behavioral: Beery- Buktenica Developmental Test of Visual Motor Integration — Investigation of visual motor integration, motor coordination and visual perception by Beery- Buktenica Developmental Test of Visual Motor Integration.
Behavioral: Jebsen Taylor Hand Function Test — Investigation of hand skills by Jebsen Taylor Hand Function Test
Diagnostic Test: Participation and Environment Measure - Children and Youth — Investigation of participation by Participation and Environment Measure - Children and Youth

SUMMARY:
The aim of this study is to compare visual-motor integration, academic achievement and participation in activities of daily living with and without type 1 diabetes.

DETAILED DESCRIPTION:
There are two different groups in this study. The first group includes children with type 1 diabetes and the second group includes healthy children. Children aged 8-12 years were included in the evaluation. Beery-Buktenica Developmental Test of Visual Motor Integration , academic achievement (Turkish, mathematics, social sciences exam scores) Participation and Environment Measure-Children an Youth, Jebsen Taylor Hand Function Test were used for evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 8 and 12,
2. To be diagnosed with Type 1 diabetes,
3. To be receiving education at primary education level,
4. Children who agree to participate in the cooperative during the evaluations,
5. Parents and children accepted to participate in the study.

Exclusion Criteria:

1. Any acute or chronic illness that affects the level of physical activity,
2. Other types of diabetes,
3. Mental problems,
4. Having received psychiatric treatment,
5. Having vision problems.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with T1DM followed in Istanbul Medipol Mega University Hospital Pediatric Endocrinology Polyclinic. Healthy children and their parents will be selected from primary and secondary schools near the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Visual Motor Integration | 30 minutes
  Visual-motor integration (VMI) is "the degree to which visual perception and finger-hand movements are well coordinated" and will asses with Beery-Buktenica Developmental Test of Visual-Motor Integration in this study. This test is a standardized, norm-referenced assessment involving copying geometric forms that is used to determine the level of integration between visual and motor systems in people of all ages. The Short Format and Full Format tests take about 10-15 minutes each to administer. Results are reported as standard scores, percentiles, and age equivalents.
Hand Skills | 10-15 minutes
  The Jebsen Taylor Hand Function Test (JTHFT) assesses both dominant and non-dominant hand skills and provides an objective assessment of hand function included in 7 subtests of daily living activities. The time (in seconds) to perform the 7 subtests is measured by the stopwatch. JTHFT is valid, reliable and normative for children.
Participation | 25-40 minutes
  Participation and Environment Measurement- Children and Youth (PEM-CY) is a parent reported measure developed in North America. Evaluates the environmental factors affecting the participation of disabled and non-disabled children and young people. It examines three environments, home, school and environment, and discusses each environment in two parts as "participation and environment".
academic achievement | 1 minutes
  Academic achievement was evaluated with Turkish, mathematics and social sciences course success points.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided